CLINICAL TRIAL: NCT05786573
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study With An Open Label Safety and Dose Confirmation Run-In Period, To Evaluate the Efficacy and Safety of Obexelimab in Patients With Warm Autoimmune Hemolytic Anemia (SApHiAre)
Brief Title: A Study of Obexelimab in Patients With Warm Autoimmune Hemolytic Anemia (SApHiAre)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zenas BioPharma (USA), LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZB012-03-002
Record Dates: First submitted 2023-03-13; First posted 2023-03-27 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Warm Autoimmune Hemolytic Anemia
Keywords: Warm Autoimmune Hemolytic Anemia; wAIHA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety and Dose Confirmation Run-in Period (SRP): Obexelimab (Experimental): Obexelimab will be administered as an SC injection for 24 weeks.
  Interventions: Drug: Obexelimab
- Randomized Control Period (RCP): Obexelimab (Experimental): Obexelimab will be administered as an SC injection for 24 weeks.
  Interventions: Drug: Obexelimab
- Randomized Control Period (RCP): Placebo (Placebo Comparator): Placebo will be administered as an SC injection for 24 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Obexelimab — Obexelimab is a monoclonal antibody that simultaneously binds CD19 and FcγRIIb, resulting in down regulation of B cell activity.
  Arms: Safety and Dose Confirmation Run-in Period (SRP): Obexelimab
Drug: Obexelimab — Obexelimab is a monoclonal antibody that simultaneously binds CD19 and FcγRIIb, resulting in down regulation of B cell activity.
  Arms: Randomized Control Period (RCP): Obexelimab
Other: Placebo — Placebo
  Arms: Randomized Control Period (RCP): Placebo

SUMMARY:
This study aims to examine the efficacy and safety of obexelimab in participants with Warm Autoimmune Hemolytic Anemia (wAIHA).

DETAILED DESCRIPTION:
This study consists of a 6-month open label Safety and Dose Confirmation Run-in Period (SRP), 6-month Randomized Control Period (RCP), and an additional 1-year open-label extension (OLE) period. To enter the Screening Period (Day -28 to Day -1) in the SRP or RCP, patients must have a clinical diagnosis of primary or secondary wAIHA due to an underlying autoimmune disorder, have failed at least 1 prior wAIHA treatment regimen, and have a Hgb level of ≥ 7 to < 10 g/dL with at least one sign or symptom of anemia. For the SRP only, patients with secondary wAIHA due to underlying lymphoproliferative disease may be eligible if they are receiving stable treatment.

All patients in the SRP or RCP are allowed to continue up to 2 failed wAIHA therapies throughout the 24-week study. On Day 1 of the SRP, patients receive obexelimab administered as subcutaneous (SC) injections. On Day 1 of the RCP, patients will be randomized in a ratio of 1:1 to receive either obexelimab or placebo administered as subcutaneous (SC) injections. Patients must return to the study site for the first 5 weeks and then every 2 weeks thereafter. Patients will undergo assessments for efficacy, safety, PK, PD, and immunogenicity during the 24-week SRP or RCP.

Following the 24-week SRP or RCP, patients will have the opportunity to receive obexelimab for up to 52 weeks in the Open Label Extension (OLE) Period.

Including screening and follow-up, the maximum duration of participation in this study for an individual patient is 81 weeks (i.e., 28-day screening, 24-week SRP or RCP, 52-week OLE, and an 8-week follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, ≥ 18 years of age
2. Clinically diagnosed with wAIHA for at least 3 months and currently receiving treatment for wAIHA or have previously received treatment for wAIHA.
3. Diagnosis of primary or secondary wAIHA documented by a positive direct antiglobulin test specific for anti-IgG or anti-IgA.
4. Failed at least 1 prior wAIHA treatment regimen.
5. At least one sign or symptom of anemia as assessed by the investigator at screening.
6. Other inclusion criteria apply.

Exclusion Criteria:

1. Have cold antibody AIHA, cold agglutinin syndrome, mixed type (i.e., warm, and cold) AIHA, or paroxysmal cold hemoglobinuria.
2. Have any other associated cause of hereditary or acquired hemolytic anemia.
3. For the RCP only, patients with secondary wAIHA not due to autoimmune disorders, including LPDs.
4. Received a transfusion within 2 weeks prior to randomization.
5. Use of B cell-depleting, B cell-targeted, or other biologic immunomodulatory agents within the 6 months prior to randomization.
6. Received IV Ig or epoetin alfa within 6 weeks prior to randomization.
7. Receiving more than 2 concomitant medications for the treatment of wAIHA.
8. Other exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Dose Confirmation Run-in Period (SRP) | 24 weeks
  Proportion of participants with hemoglobin (Hgb) ≥ 10 g/dL and ≥ 2 g/dL increase from Baseline with no use of blood transfusion or glucocorticoid (GC) rescue therapy.
Randomized Control Period (RCP) | 24 weeks
  Proportion of participants who achieve a durable Hgb response (defined as Hgb ≥ 10 g/dL and ≥ 2 g/dL increase from Baseline on at least 3 of 4 consecutive available visits), at the earliest on or after Week 12, with no use of blood transfusion or GC rescue therapy prior to attaining durable response through Week 24.

CONTACTS AND LOCATIONS:
Locations (7):
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
- Copernicus PL Sp. z o.o. Wojewodzkie Centrum Onkologii, Gdansk, Pomeranian Voivodeship, Poland
- Spain (2):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario 12 de Octubre, Madrid
- National Cheng Kung University Hospital, Tainan, Taiwan
- United Kingdom (2):
  - Plymouth Hospitals NHS Trust, Plymouth, Devon
  - Kent and Canterbury Hospital, Canterbury, Kent